CLINICAL TRIAL: NCT03173391
Title: A 24-week Multi-center, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of HMS5552 With Additional 28-week Open-label Treatment to Evaluate the Safety of HMS5552 Alone in T2DM Subjects
Brief Title: Long-term Efficacy and Safety of HMS5552 in T2DM Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMM0301
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GKA; T2DM; HMS5552; monotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin; glucokinase activator compound 50

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMS5552 (Experimental): 75mg BID
  Interventions: Drug: HMS5552
- Placebo (Placebo Comparator): BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMS5552 — BID Oral administration
  Other Names: Glucokinase Activator (GKA)
  Arms: HMS5552
Drug: Placebo — BID Oral administration
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety and population PK of HMS5552 as monotherapy in adult type 2 diabetic subjects, there will be 2 groups in the first 24 weeks, one group will receive HMS5552 , while the other group will receive placebo ; after 24 weeks, all subjects will receive HMS5552 for 28 weeks.

DETAILED DESCRIPTION:
This study is a phase III study in subjects with T2DM. As designed, the study will start with a 4-week, single-blind, placebo run-in period based on diet and exercise interventions for screening eligible subjects. The eligible subjects are randomly assigned to HMS5552 75mg BID group or placebo BID group with ratio 2:1 to receive a 24-week double-blind treatment. Then all subjects receive 28-week open-label treatment of HMS5552 75mg BID . After 52-week treatment, all investigational drugs should be discontinued, followed by 1 week for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18~75 years old
2. naive T2DM 3.7.5% ≤ HbA1c ≤ 11.0% at screening 4.18.5 kg/m2 < BMI < 35.0 kg/m2 at screening;

Exclusion Criteria:

1. T1DM
2. Fasting C-peptide <1.0 ng/ml (0.33 nmol/L) at screening
3. Medical history of severe hypoglycemia, diabetic ketoacidosis, diabetes lactic acidosis or hyperosmotic nonketotic diabetic coma, severe cardio-cerebrovascular,unstable or rapidly progressive kidney disease, active liver diseases,diagnosed mental disease,etc

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | 24 weeks
  The change of HbA1c from baseline in T2DM subjects after 24-week double-blind treatment

SECONDARY OUTCOMES:
The change of 2-hour postprandial plasma glucose (2h-PPG) from baseline | 24 weeks
  The change of 2-hour postprandial plasma glucose (2h-PPG) from baseline in T2DM subjects after 24-week double-blind treatment
The change of fasting plasma glucose (FPG) from baseline | 24 weeks
  The change of fasting plasma glucose (FPG) from baseline in T2DM subjects after 24-week double-blind treatment
The proportion of subjects with HbA1c < 7.0% | 24 weeks
  The HbA1c response rate in T2DM subjects after 24-week double-blind treatment
Incidence of Treatment-Emergent Adverse Events over time | 52 weeks
  including incidence of adverse events, incidence of hypoglycemic events, physical examination, vital signs, 12-lead ECG, clinical laboratory examinations (routine blood test, blood biochemistry and routine urine test).

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Hua Medicine Limited, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No